CLINICAL TRIAL: NCT03588988
Title: Effect of Dexmedetomidine on Postoperative Delirium Inflammasome Activation Inhibition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2018-0472
Record Dates: First submitted 2018-07-03; First posted 2018-07-17 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Patients Under Hip, Femur, Spine Operation
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental)
  Interventions: Drug: Dexmedetomidine IV infusion
- Control group (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine IV infusion — Patients who underwent spine, hip or femur surgery and who were admitted to the ICU after institutional exhalation were randomly assigned to the DEX group and the control group. Both groups can be combined with remifentanil for appropriate postoperative analgesia. The DEX group injects DEX at 0.2 ug / kg / hr from 9 pm to 7 am. At this time, the patient's blood pressure, oxygen saturation and cardiopulmonary function are continuously monitored.
  Arms: Dexmedetomidine group
Drug: Normal saline — Patients who underwent spine, hip or femur surgery and who were admitted to the ICU after institutional exhalation were randomly assigned to the DEX group and the control group. Both groups can be combined with remifentanil for appropriate postoperative analgesia. The control group is inoculated with saline solution. At this time, the patient's blood pressure, oxygen saturation and cardiopulmonary function are continuously monitored.
  Arms: Control group

SUMMARY:
Delirium is an acute or subacute comorbid syndrome characterized by decreased awareness and cognitive dysfunction accompanied by attention deficit. It varies from 20% to 80%, depending on the report. If delirium occurs in intensive care unit, complications such as intubation tube and catheter removal that are not desired are increased, mechanical ventilation deviation is prolonged, and eventually the intensive care unit is extended. Prevention of delirium is therefore very important, but no medication has been found to prevent delirium.

Recent studies have shown that pro-inflammatory cytokines play an important role in the development of delirium, and as a result of the stimulation of the peripheral inflammatory reaction, proinflammatory cytokines (interleukin (IL) -6, tumor necrosis factor- ), And IL-10) secretion, resulting in the induction of inflammatory responses of the central nervous system. In addition, sleep habits have been shown to affect the pro-inflammatory pathway, and sleep induction and inactivation of the pro-inflammatory pathway may be expected to prevent and treat delirium.

Dexmedetomidine (DEX) is a highly selective a2-agonist with sedative and analgesic effects and reduces sympathetic response to stimuli. Compared to benzodiazepine and opioid, there are fewer side effects of respiratory depression.

In animal studies, the possibility of intrinsic immune suppression of DEX has been demonstrated, and recent studies have shown that intravenous DEX administration reduces IL-6, IL-8, and TNF-a levels, resulting in anti-inflammatory effects. IL-6 plays a key role in neuroinflammation with both proinflammatory cytokines and anti-inflammatory cytokines, including infection, traumatic brain injury, ischemia, and neurodegenerative disorders. DEX plays a key role in IL-6 stimulated IL-6 And inhibits mRNA expression and thus has a brain function-protecting effect. In clinical trials, DEX administration compared with propofol decreased IL-6 secretion and decreased post-operative cognitive impairment in ICU patients after primary surgery. This is closely related to the formation of inflammatory complexes (Inflammasome). In addition, low-dose DEX infusion in patients with ICU at night has a low incidence of delirium during the ICU period, and studies have shown that sleep quality is improved in the DEX group in the mechanical ventilation group. Patients who did not undergo mechanical ventilation also reported improved sleep quality with prophylactic low-dose DEX. As such, the definitive mechanism has not yet been clarified, but the use of low-dose DEX is increasingly proactively used to improve sleep quality.

The purpose of this study was to investigate the effect of DEX on the inflammatory pathway during nighttime after ICU admission and to observe the quality of sleep and the prognosis of delirium.

DETAILED DESCRIPTION:
Delirium is an acute and subacute comorbid syndrome characterized by decreased awareness and cognitive dysfunction accompanied by attention deficit. It varies from 20% to 80% in patients entering the ICU. If delirium occurs in the intensive care unit, complications such as unintended intubation, unintentional drainage, and mechanical ventilation are prolonged. Prevention of delirium is therefore very important, but no medication has been found to prevent delirium. Recent studies have shown that the pro-inflammatory cytokine affects the etiology of delirium. In addition, sleep habits have been shown to affect the pro-inflammatory pathway, and sleep induction and inactivation of the pro-inflammatory pathway may be expected to prevent and treat delirium.

DEX is a selective alpha-2 receptor agonist with sedative and anti-anxiety effects and reduces sympathetic response due to stimulation. Recent studies have shown that intravenous DEX is effective in reducing inflammation by decreasing levels of IL-6, IL-8, and TNF-a.

This study investigated the effect of dexmedetomidine, which is continuously administered at night after ICU admission, on the development of delirium and inflammatory markers, and to observe the prognosis. Patients who underwent spine, hip or femur surgery and who were admitted to the ICU after institutional exhalation were randomly assigned to the DEX group and the control group. Both groups can be combined with remifentanil for appropriate postoperative analgesia. The DEX group injects DEX at 0.2 ug / kg / hr from 9 pm to 7 am. The control group is inoculated with saline solution. At this time, the patient's blood pressure, oxygen saturation and cardiopulmonary function are continuously monitored. If an adverse event occurs during DEX sedation, process it and record it. If hypotension occurs, 4 mg of IV ephedrine is administered. If hypotension occurs, 4 mg is added or infused with norepinephrine. If Bradycardia (HR <45 bpm) occurs, IV glycopyrrolate 0.2 mg is administered. If bradycardia persists after administration, administer 0.5 mg IV atropine at a maximum of 0.5 mg. If respiratory depression (RR <10 / min) and hypoxia (SaO2 <90%) occur, the patient may be awakened by loud or mild stimulation. If the respiratory depression and hypoxia persist despite these treatments, head extension , and maneuver for airway maintenance such as jaw thrust.

IL-1β, IL-6, TNF-α, caspase-1, NLRP3 and ASC were measured at the onset of surgery in both the DEX group and the control group. Follow up.

The following morning the subjects themselves and the researchers evaluate the quality of sleep (using RCSQ questionnaire) and delirium (ICDSC, CAM-ICU), respectively.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I to III adults
* aged 20 years or older who can read and understand the consent form
* patients who have been admitted to the ICU after institution of hip, femur, and spine surgery

Exclusion Criteria:

* Patients who do not understand and understand the written consent of an illiterate or foreigner
* pregnant woman
* 20 years old
* Patients with moderate to severe liver disease (AST, ALT> 200 IU / L)
* Patients with end stage renal disease (eGFR <30 or dialysis patients)
* allergy to DEX, presence of electrocardiographic atrioventricular block, hemodynamic instability
* Left ventricular ejection fraction <30%, congestive heart failure, severe coronary artery disease, hemodynamically unstable arrhythmia

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
CRP(C-reactive protein) | Post operative day 0
  Effect of dexmedetomidine(DEX) on post-conditioning delirium and inflammasome activation
CRP(C-reactive protein) | Post operative day 1
  Effect of dexmedetomidine(DEX) on post-conditioning delirium and inflammasome activation
the number of Neutrophil or Lymphocyte | Post operative day 0
  Effect of dexmedetomidine(DEX) on post-conditioning delirium and inflammasome activation
the number of Neutrophil or Lymphocyte | Post operative day 1
  Effect of dexmedetomidine(DEX) on post-conditioning delirium and inflammasome activation
total score of Richards-Campbell Sleep Questionnaire(RCSQ) obtained by summing each score out of 100 | Post operative day 0
  double-checked RCSQ; one is patient check, and the other is night nurse check.
total score of Richards-Campbell Sleep Questionnaire(RCSQ) obtained by summing each score out of 100 | Post operative day 1
  double-checked RCSQ; one is patient check, and the other is night nurse check.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No